CLINICAL TRIAL: NCT06754995
Title: Diagnostic Feasibility of 100 Hz Tetanic Stimulation in the Perioperative Setting in Patients With Normal and Abnormal ENG: a Pilot Study
Brief Title: Diagnostic Feasibility of 100 Hz Tetanic Stimulation
Status: Recruiting | Type: Observational
Sponsor: University of Debrecen (Other)
Responsible Party: Principal Investigator, Pongrácz Adrienn, assistant professor, University of Debrecen
Other Study IDs: AITT 2024/2
Record Dates: First submitted 2024-12-05; First posted 2025-01-01 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-12

CONDITIONS: Polyneuropathies
Keywords: electromyography; electroneurography; tetanic stimulation; residual neuromuscular block; neuromuscular monitoring
MeSH Terms: conditions — Polyneuropathies; Delayed Emergence from Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Normal ENG: Patients who have normal results at baseline electroneurogrphy examination
- Abnormal ENG: Patients who have abnormal results at baseline electroneurogrphy examination due to polyneuropathy

SUMMARY:
The goal of this observational study is to investigate the applicability of 100 Hz tetanic stimulation with an electromyography device in the exclusion of postoperative residual neuromuscular block. The aim is to determine whether fatigue develops with 100 Hz tetanic stimulation in anaesthetized, non-relaxed patients with normal or abnormal baseline electroneurographic (ENG) findings.

DETAILED DESCRIPTION:
The aim of the present study is to investigate the applicability of 100 Hz tetanic stimulation with an electromyography (EMG) device. The aim is to determine whether fatigue develops with 100 Hz tetanic stimulation in anaesthetized, non-relaxed patients with normal or abnormal baseline electroneurographic (ENG) findings. Electric responses of the musculus digiti minimi elicited by supramaximal stimulation of the ulnar nerve at the carpal tunnel are monitored. Alpine Biomed ENG-EMG device with Keypoint software version 5.11 is used for the examinations. The exposed arm is fixed on the armboard, the skin is degreased and then the electrodes for monitoring are mounted lege artis. After the anesthesia has been induced, ENG of the ulnar nerve is examined. Based on the results of the ENG test, patients are divided into separate groups (normal or abnormal ENG). During the ENG test, the supramaximal current is determined. Afterwards, repetitive tetanic stimulation of the defined frequency (60 and 100 Hz) and duration (5 sec) is applied to the two test groups at the current according to the test plan.

The clinical utilities of the study results are:

* Determination of the "safety margin" of neuromuscular junction, which is not provided by routine monitoring.
* To investigate how comorbid status (especially chronic conditions affecting peripheral nerves such as polyneuropathy) influences the feasibility of tetanic stimulation in the diagnostics of residual neuromuscular block and safety margin.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3;
* BMI 18.5-25 (normal body weight);
* patient is in supine position with one arm accessible.

Exclusion Criteria:

* diseases with impaired neuromuscular function (myopathies, severe liver and kidney failure);
* drugs affecting neuromuscular function (magnesium, aminoglycosides);
* pregnancy (pregnancy tests are carried out in women of childbearing age to rule out pregnancy);
* breast-feeding;
* acute surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgical patients
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-01-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
100 Hz tetanic fade response of abductor digiti minimi muscle to ulnar nerve stimulation in patients with normal and abnormal ENG | From enrollment until end of anesthesia asessed up to 1 hour. No further ENG measurements are performed in the postoperative period.
  Electroneurography response of the abductor digiti minimi muscle to 100 Hz tetanic stimulation (tetanic fade) is examined to find out if there is difference in patients with or without polyneuropathy. Tetanic fade is the decrease of the twitch heights of the compound muscle action potential due to depletion of cetylcholin stores in the nerve terminal during tetanic stimulation.

SECONDARY OUTCOMES:
Diagnostic feasibility of electromyography in the examination of safety margin | From enrollment until end of anesthesia assessed up to 1 hour. No further ENG measurements are performed in the postoperative period.
  To see whether tetanic stimulation with electromyography can be used as a routine tool to examine the safety margin and residual neuromuscular block. It is expected that there will be no fade in muscle response to 60 Hz tetanic stimulation in either groups. It is suspected that there will be no tetanic fade response to 100 Hz tetanic stimulation in patinets with normal ENG, however patinets with abnormal baseline ENG will produce tetanic fade. The incidence and extent of tetanic fade response will be examined.

OTHER OUTCOMES:
60 Hz tetanic fade response of abductor digiti minimi muscle to ulnar nerve stimulation in patients with normal and abnormal ENG | From enrollment until end of anesthesia assessed up to 1 hour. No further ENG measurements are performed in the postoperative period.
  Electroneurography response of the abductor digiti minimi muscle to 60 Hz tetanic stimulation (tetanic fade) is examined to find out if there is difference in patients with or without polyneuropathy. Tetanic fade is the decrease of the twitch heights of the compound muscle action potential due to depletion of cetylcholin stores in the nerve terminal during tetanic stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Béla Fülesdi, MD PhD DSci, Study Director — University of Debrecen
Locations (2):
- Hungary (2):
  - Department of Anesthesiology and Intensive Care, University of Debrecen, Debrecen, Hajdú-Bihar
  - University of Debrecen Medical Center, Department of Anesthesiology and Intensive Care, Debrecen

IPD SHARING:
Plan to Share IPD: No